CLINICAL TRIAL: NCT06944444
Title: A Phase I Clinical Study of the Safety, Pharmacokinetics, and Antitumor Activity of SSS59 in Patients With Advanced Malignant Tumors
Brief Title: A Phase I Clinical Study of SSS59 Monotherapy in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSS59-101
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A1 (Experimental): Dose escalation will be conducted using accelerated titration and traditional 3+3 design. Dose Escalation Level includes 12 levels, QW IV. Dose extension will be carried out at the selected level.
  Interventions: Drug: SSS59
- Part A2 (Experimental): Dose escalation will be conducted using a traditional 3+3 design. Dose Escalation Level includes 12 levels, Q2W IV. Dose extension will be carried out at the selected level.
  Interventions: Drug: SSS59
- Part A3 (Experimental): Dose extension will be carried out at the selected dose level, Q3W, IV.
  Interventions: Drug: SSS59
- Part B (Experimental): Indication extension will be carried out at the selected level.
  Interventions: Drug: SSS59

INTERVENTIONS:
Drug: SSS59 — A humanized antibody targeting MUC17

SUMMARY:
This study was an open-label phase I study to evaluate the safety, pharmacokinetics, and antitumor activity of SSS59 as a single agent in patients with advanced malignancies.

DETAILED DESCRIPTION:
This study includes 4 Parts: Part A1 (dose escalation and dose extension for QW administration), Part A2 (dose escalation and dose extension for Q2W administration), Part A3 (dose extension for Q3W administration), and Part B (indication extension, such as advanced gastric or gastroesophageal junction adenocarcinoma with MUC17 positive, failure of standard therapy, or intolerance to standard therapy , or other tumors).

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically documented local advanced or recurrent or metastatic malignancies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival >3 months.
* Signed informed consent form.
* Must have adequate organ function.

Exclusion Criteria:

* Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5. 0, with exception of hair loss and fatigue.
* Pregnant or nursing women or women/men who are ready to give birth.
* symptomatic central nervous system metastasis.
* Allergy to other antibody drugs or any excipients in the study drugs.
* Underwent major surgery within 4 weeks prior to first dosing.
* The patient is participating in another clinical study, unless it is an observational (non-intervention) clinical study or a follow-up period of an intervention study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DLTs | 21 days
  Dose limiting toxicity
Safety and tolerability | during the intervention，Within 28 days of the last dose
  Safety and tolerability assessed by incidence and severity of adverse events
MTD and RP2D | through study completion, an average of 2 year
  Determine the maximum tolerated dose and determine the recommended phase II dose

SECONDARY OUTCOMES:
Cmax of SSS59 | baseline, during the intervention and at the end of the study
  Maximum concentration
Tmax of SSS59 | baseline, during the intervention and at the end of the study
  Time to peak drug concentration
AUC0-last of SSS59 | baseline, during the intervention and at the end of the study
  the area under the curve (AUC) up to the last measurable concentration
RO of SSS59 | baseline, during the intervention and at the end of the study
  Receptor Occupancy
Pharmacodynamic (PD) characteristics of SSS59 | baseline, during the intervention and at the end of the study
  change of cytokine
Immunogenicity of SSS59 | baseline, during the intervention and at the end of the study
  ADA，NAB（if ADA is positive）
Preliminary antitumor activity of SSS59 | baseline, during the intervention and at the end of the study
  Assessed according to Recist V1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No